CLINICAL TRIAL: NCT00273377
Title: The Effects of Hypercapnia, Supplemental Oxygen, and Dexamethasone on Surgical Wound Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 302; NIH Grant GM 061655; Gheens Foundation; Joseph Drown Foundation
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Surgical Wound Infection; Surgery, Colon
Keywords: Anesthesia; Oxygen; Carbon dioxide; Hypercapnia; Hypercarbia; Dexamethasone; Steroid; Postoperative nausea and vomiting (PONV)
MeSH Terms: conditions — Surgical Wound Infection; Hypercapnia; Postoperative Nausea and Vomiting | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Mild intraoperative hypercapnia (50 mmHg vs. 30 mmHg)
Other: Supplemental oxygen (80% vs. 30%)
Drug: Dexamethasone — 4 mg
Drug: Placebo — placebo

SUMMARY:
The investigators will test the hypotheses that mild hypercapnia and supplemental oxygen reduce wound infection risk in patients undergoing colon resection. The investigators will simultaneously test the hypothesis that low-dose dexamethasone (a common treatment for postoperative nausea and vomiting) does not increase infection risk.

DETAILED DESCRIPTION:
Wound infections are common and serious complications of anesthesia and surgery. Even in patients who are kept normothermic and given supplemental oxygen, the incidence of wound infection after colon resection exceeds 5%. About 80% of these resections are done for colon cancer, the third leading cause of cancer death. The average surgical wound infection prolongs hospitalization by a week and substantially increases cost. Major factors influencing the incidence of surgical wound infection include the site and complexity of surgery, underlying illness (including treatment with immunosuppressive drugs), timely administration of prophylactic antibiotics, intraoperative patient temperature, hypovolemia, and tissue oxygen tension.

The primary defense against surgical pathogens is oxidative killing by neutrophils. Oxygen is a substrate for this process, and the reaction critically depends on tissue oxygen tension throughout the observed physiological range. It is therefore unsurprising that subcutaneous tissue oxygen tension (PsqO2) is inversely correlated with the risk of surgical wound infection. Primary determinants of tissue oxygen availability include arterial oxygen tension, hemoglobin concentration, and local perfusion.

An additional determinant of peripheral oxygen delivery is cardiac output. Mild hypercapnia increases cardiac output: for example, augmenting arterial carbon dioxide tension (PaCO2) just 10-12 mmHg increases the cardiac index 15%. Our preliminary studies confirm that mild hypercapnia increases cardiac output and additionally indicate the hypercapnia markedly improves tissue oxygenation. For example, tissue oxygen tension increased 16 mmHg, from 58 to 74 mmHg over a 20 mmHg range of PaCO2 in anesthetized volunteers. We have also shown that increasing PaCO2 by just 15 mmHg increased tissue oxygen tension 16 mmHg in surgical patients. Similar results were observed in morbidly obese patients. Previous work indicates that similar increases in PsqO2 reduces the risk of surgical wound infection by about 30%. We thus propose to test the hypothesis that mild hypercapnia significantly reduces the incidence of surgical wound infection in normothermic patients undergoing colon resection. Secondary outcomes will include the duration of hospitalization, cost of care, the incidence of nosocomial pneumonia, the incidence of postoperative nausea and vomiting (PONV) and return to function.

High intra- and postoperative oxygen concentration (80%, as opposed to 30% oxygen) has been shown to reduce the rate of wound infection by more than 50%. Therefore, the protocol implemented high intraoperative oxygen concentrations for all patients this trial. However, within the first 500 enrolled patients a recent trial reported a better outcome for patients with low perioperative oxygen concentrations. Although that trial was less well controlled and underpowered, the conflicting evidence indicates that additional study is needed. We will therefore simultaneously test the hypothesis that supplemental oxygen reduces infection risk.

Patients undergoing colon surgery are generally at high risk for postoperative nausea and vomiting (PONV). According to results from meta-analyses, a single intraoperative dose of dexamethasone is effective and safe for the prophylaxis for PONV. Dexamethasone has thus been recommended as a first-line prophylaxis for PONV. However, none of the previous PONV trials have focused on wound infections nor had a sufficiently long observational period to rule out potential concerns of an increased incidence of wound infection. We will therefore also test the hypothesis that dexamethasone does not increase the risk of surgical wound infection. The second and third hypotheses will be added to the protocol, using a factorial design, after the first 500 patients are enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Colon resection expected to last >2 and <6 hours

Exclusion Criteria:

* Bowel obstruction
* Fever

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2002-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Surgical wound infection | 30 days

SECONDARY OUTCOMES:
Duration of hospitalization | 30 days
Suture removal | 30 days
Cost of care | 30 days
Return to work | 30 days
Nosocomial pneumonia | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, M.D., Study Director — The Cleveland Clinic; Ozan Akca, M.D., Principal Investigator — University of Louisville
Locations (4):
- United States (2):
  - Outcomes Research Institute, Louisville, Kentucky
  - Cleveland Clinic, Cleveland, Ohio
- University of Vienna, Vienna, Austria
- Mater Misericordiae Hospital, Dublin, Ireland

REFERENCES:
- [Derived] Kurz A, Fleischmann E, Sessler DI, Buggy DJ, Apfel C, Akca O; Factorial Trial Investigators. Effects of supplemental oxygen and dexamethasone on surgical site infection: a factorial randomized trialdouble dagger. Br J Anaesth. 2015 Sep;115(3):434-43. doi: 10.1093/bja/aev062. Epub 2015 Apr 20. PMID 25900659
- [Derived] Akca O, Kurz A, Fleischmann E, Buggy D, Herbst F, Stocchi L, Galandiuk S, Iscoe S, Fisher J, Apfel CC, Sessler DI; Hypercapnia Trial Investigators. Hypercapnia and surgical site infection: a randomized trial. Br J Anaesth. 2013 Nov;111(5):759-67. doi: 10.1093/bja/aet233. Epub 2013 Jul 24. PMID 23887247